CLINICAL TRIAL: NCT02129426
Title: Comparison of Outcomes During MRI Sedation With Midazolam-dexmedetomidine Versus Ketamine-dexmedetomidine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit the adequate number of subjects
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, John W Berkenbosch, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Ket-Dex/M-Dex MRI
Record Dates: First submitted 2014-04-23; First posted 2014-05-02 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Sedation
Keywords: Sedation; MRI
MeSH Terms: interventions — Ketamine; Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine and Ketamine (Experimental): Subjects will already be getting Dexmedetomidine and Ketamine for their routine care.
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine
- Dexmedetomidine and Midazolam (Active Comparator): Subjects will already be getting Dexmedetomidine and Midazolam for their routine care.
  Interventions: Drug: Midazolam; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketamine — Sedation medication
  Arms: Dexmedetomidine and Ketamine
Drug: Midazolam — Sedation medication
  Arms: Dexmedetomidine and Midazolam
Drug: Dexmedetomidine — Sedation medication

SUMMARY:
This study will compare 2 different sedation drugs (Ketamine and Midazolam) when they are used with another sedating medicine called Dexmedetomidine for MRI sedation. This study hopes to measure the impact each drug has on what happens during and after MRI sedation with Dexmedetomidine

DETAILED DESCRIPTION:
The will be a randomized, double-blind, prospective study. All patients referred to UCSS for brain MRI and for whom dexmedetomidine would otherwise be the sedation regimen of choice will be eligible for enrollment. The investigators propose to limit the study to patients undergoing only brain MRI as these studies are of a predictable length (25-30 minutes); therefore the sedation regimen can be more easily standardized. Parents of eligible patients would be approached prior to or during the pre-sedation assessment and told about the study and, if they agree to enroll, informed consent would be obtained. Assent will be obtained from children 7 years of age and greater, if they are otherwise developmentally capable of giving assent. The goal is to enroll 50 subjects (25 per treatment group) which would be sufficient to detect a 25% or greater difference in the mean maximal heart rate or blood pressure decrease from baseline between the 2 groups.

Following consent, subjects would be randomized to be sedated with either midazolam-dexmedetomidine or ketamine-dexmedetomidine and, upon achieving an appropriate depth of sedation, undergo their MRI. Monitoring during the MRI and subsequent recovery would occur in compliance with the current Norton Children's Hospital Sedation policy. Recovery-related behavior would be assessed using the Pediatric Anesthesia Emergence Delirium Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient at Kosair Children's Hospital.
2. Order placed by treating team for MRI of the brain with sedation.
3. Age less than or equal to 18 years.
4. Plan to sedate with dexmedetomidine, regardless of study participation.

Exclusion Criteria:

1. Previous adverse reaction to dexmedetomidine or clonidine
2. Current use of clonidine as a routine medication
3. Concurrent use of a heart-rate decreasing medication (digoxin, propranolol)
4. Contraindication to ketamine use

   * Intracranial hypertension or traumatic brain injury
   * Intraocular hypertension of eye trauma
   * Pulmonary hypertension requiring medical management
5. Planned additional procedure during the sedation encounter (non-brain MRI, lumbar puncture, EEG etc)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Berkenbosch, M.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine and Ketamine: Subjects will already be getting Dexmedetomidine and Ketamine for their routine care.
  Ketamine
  Dexmedetomidine
- Dexmedetomidine and Midazolam: Subjects will already be getting Dexmedetomidine and Midazolam for their routine care.
  Midazolam
  Dexmedetomidine
Period: Overall Study
Arm/Group | Dexmedetomidine and Ketamine | Dexmedetomidine and Midazolam
Started | 7 | 13
Completed | 0 | 0
Not Completed | 7 | 13

BASELINE CHARACTERISTICS:
Population: 21 subjects enrolled however, 1 subject's data was on paper archived and not available to perform demographic analysis therefore is not included here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine and Ketamine | Dexmedetomidine and Midazolam | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 13 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] — Collected: age and sex, weight, BMI, primary diagnosis, and reason for MRI race/ethnicity not collected per protocol
  months | 27 (23) | 35 (18) | 32.2 (19.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data was not collected.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 13 | 20
BMI [Mean (Standard Deviation); unit: kilogram per meter squared] | 16.4 (1.5) | 17.4 (2.6) | 17.0 (2.2)
Primary Diagnosis [Number; unit: participants]
  seizure | 7 | 7 | 14
  Diplopia | 0 | 1 | 1
  Ataxia | 0 | 4 | 4
  syncope | 0 | 1 | 1
MRI Indication [Count of Participants; unit: Participants]
  Seizure | 7 | 7 | 14
  Diplopia | 0 | 1 | 1
  Ataxia | 0 | 4 | 4
  Syncope | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Hypotension and/or Bradycardia During Sedation and Recovery (Generally 2-3 Hours)
Description: number of participants developing hypotension and or bradycardia
Time Frame: a total of 2-3 hours during sedation and recovery.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine and Ketamine | Dexmedetomidine and Midazolam
Number analyzed (Participants) | 7 | 13
Participants
  Hypotension | 0 | 0
  Bradycardia | 0 | 0

2. Secondary Outcome: Percent Change in Heart Rate From Baseline
Description: Change in heart rate from baseline.
Time Frame: during sedation and recovery (generally 2-3 hours)
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Dexmedetomidine and Ketamine | Dexmedetomidine and Midazolam
Number analyzed (Participants) | 7 | 13
percent change from baseline | -29.9 (7.5) | -29.6 (11.1)
Statistical Analysis 1: Comparison: Dexmedetomidine and Ketamine vs Dexmedetomidine and Midazolam; Test type: Other — t-test comparison of the two groups; p = 0.96, t-test, 1 sided

3. Secondary Outcome: Percent Change in Blood Pressure From Baseline
Description: Change in blood pressure from baseline.
Time Frame: during sedation and recovery (generally 2-3 hours)
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Dexmedetomidine and Ketamine | Dexmedetomidine and Midazolam
Number analyzed (Participants) | 7 | 13
percent change from baseline | -18.7 (12.2) | -14.9 (11.8)
Statistical Analysis 1: Comparison: Dexmedetomidine and Ketamine vs Dexmedetomidine and Midazolam; Test type: Other; p = 0.52, t-test, 1 sided

4. Secondary Outcome: The Number of Participants With Adverse Recovery-related Behaviors During Sedation Recovery
Description: This study will compare the number of participants with adverse recovery-related behaviors, based on the PAED scores, between the 2 treatment arms.
Time Frame: Recovery-related behaviors will be specifically measured using the "Pediatric Anesthesia Emergence Delirium (PAED)" scale every 5 minutes from procedure completion until sedation recovery is complete (usually less than 2 hrs)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine and Ketamine | Dexmedetomidine and Midazolam
Number analyzed (Participants) | 7 | 13
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Dexmedetomidine and Ketamine | Dexmedetomidine and Midazolam
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 0/7 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT02129426/Prot_SAP_000.pdf